CLINICAL TRIAL: NCT02765425
Title: Training the Brain with a Robotic Device for Balance Recovery in Near-frail Older Adults
Brief Title: Training the Brain with a Robotic Device for Balance Recovery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of department staff and COVID
Sponsor: University of Arkansas (Other)
Collaborators: AMES Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 204820
Record Dates: First submitted 2016-04-07; First posted 2016-05-06 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2020-11

CONDITIONS: Fall Risk; Healthy Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Training Group (Experimental): Subjects will receive the same outcome measures at baseline, after 3 months training and 6 months later. Intervention will comprise of three sessions seated at the AMES device. Each training session will include 15 min of training of each ankle. Training sessions will be conducted 3 times/week over a 12-week period, for a total of 9 hours of training on each ankle.
  Interventions: Device: AMES
- Control Group (No Intervention): Subjects will receive no intervention. Subjects will receive all outcome measures at baseline and at 3 months post enrollment. Subjects will also receive a fall-incidence reporting form 9 months post enrollment. No other intervention - i.e. no treatment - is given.

INTERVENTIONS:
Device: AMES — Subjects will be trained while seated on the AMES device. As the footplate of the device rotates the ankle ±15 deg in dorsiflexion and plantarflexion, the participant will assist that motion. Vibration (2-3 mm at 60 pulses/s) will be applied to the tibialis anterior tendon during plantarflexion and to the Achilles tendon during dorsiflexion. To assist participants in the assisted movement task, the AMES biofeedback screen will provide real-time visual feedback of the volitional ankle torque that the participants actively apply to the AMES device. Each training session will include 15 min of training of each ankle; training sessions will be conducted 3 times/week over a 12-week period, for a total of 9 hours of training on each ankle.
  Arms: Training Group

SUMMARY:
The research objective of this study is to determine whether an intervention and associated robotic device called "Assisted Movement with Enhanced Sensation (AMES) can be used to enhance balance recovery following an unexpected loss of balance by conditioning areas of the brain involved in lower-limb (LL) motor control. It is hypothesized that AMES can improve balance recovery, gait, and reduce falls in near-frail elderly people by improving LL strength, speed, and coordination.

AMES, is a medical intervention and robotic device originally developed to aid patients' recovery from injuries to the central nervous system that limit movement. Earlier published studies demonstrated a unique property of AMES, namely that it is capable of reducing sensorimotor impairment in the severely impaired, an underserved population of patients with brain and spinal cord injuries. AMES applies assisted movement, biofeedback, and sensory stimulation simultaneously and non-invasively to the upper or lower limb, the initial intent being to address impairments such as weakness, spasticity, sensory loss, and dyssynergia (i.e., co-contraction). These reductions in impairment are achieved through cortical plasticity. In the present study, the same methodology will be applied to the lower limbs of the near-frail elderly to reduce falls by training faster reaction times, stronger reactions, and more coordinated recoveries from slips and trips

DETAILED DESCRIPTION:
The specific aim of this study is to determine preliminarily the efficacy of the AMES intervention in helping older adults quickly readjust their posture in order to recover from unexpected loss of equilibrium. An AMES device will be placed into operation at the University of Arkansas for Medical Sciences (UAMS) Out-patient Rehabilitation Therapy Clinic at Fayetteville, Arkansas(AR), where we will recruit 20 healthy, but near-frail subjects. Ten of these participants will be randomly assigned to a treatment group, and the other 10 will be assigned into a control group that will not receive the AMES intervention. Before and after 12 weeks of training with the bipedal AMES device, ankle strength, range of motion, proprioception, and reaction time, as well as gait and whole-body stability following unexpected balance perturbations will be assessed. In addition to measuring sensorimotor impairment and static balance equilibrium,the incidence of falls in all 20 participants beginning with enrollment into the study for a total of 6 months will be tracked. A reduction in sensorimotor impairment, an improvement in dynamic balance, and a reduction in fall incidence in the treatment group, but not in the control group is expected.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 65 years to 90 years old, inclusive
* With a history of one or more falls in the last 2 years
* Able to independently ambulate
* Ability to fit the legs into the AMES device
* Cognitively able to comply with instructions

Exclusion Criteria:

* Presence of substantial somatosensory deficits in the legs (i.e., <70% correct on the Joint Position Test)
* Co-morbidities that affect the ability to exercise or move the legs
* Significant history of cardiac or peripheral vascular problems that would preclude seated ankle exercises
* Participation in any other concurrent study involving the LL
* Initiation of any considered new exercise or therapeutic regimens during the study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-09-09 (Estimated); Study Completion 2020-09-09 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Falls | Prior to training (baseline) and after 3 months training
  Fall Incidence Questionnaire that records the self-reported number and type of falls.

SECONDARY OUTCOMES:
ABC Fear of Falling Questionnaire | Prior to training (baseline) and again after 3 months training
  The Activities-specific Balance Confidence (ABC) Scale is a 16-item self-report measure in which subjects rate their balance confidence for performing activities. This stem is used to lead into each activity considered: "How confident are you that you will not lose your balance or become unsteady when you..." Items are rated on a rating scale that ranges from 0 - 100 Score of zero represents no confidence, a score of 100 represents complete confidence Overall score is calculated by adding item scores and then dividing by the total number of items.

CONTACTS AND LOCATIONS:
Overall Officials: John R Jefferson, PhD, PT, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No